CLINICAL TRIAL: NCT01988701
Title: Lymphocyte Profiles and Activation Status in the Development of Chronic Graft-versus-Host Disease
Brief Title: Lymphocyte Profiles and Activation Status in Patients With Graft-Versus-Host Disease
Status: Withdrawn | Type: Observational
Why Stopped: Decision made by the PI to withdraw study
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Samantha Jaglowski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-12208; NCI-2013-01641 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Graft Versus Host Disease; Hematopoietic/Lymphoid Cancer
Keywords: GVHD; chronic Graft versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Allogeneic SCT Groups: Patients who have received stem cell transplantation at The Ohio State University are eligible and who are at or beyond day +75 following allogeneic SCT regardless of previous diagnosis of acute or chronic GVHD.
  Interventions: Other: Ancillary-Correlative
- Autologous SCT group: Patients who have received an autologous stem cell transplant at The Ohio State University and who have achieved platelet and neutrophil engraftment.
  Interventions: Other: Ancillary-Correlative

INTERVENTIONS:
Other: Ancillary-Correlative — Blood samples are analyzed for activation status of B lymphocytes, T lymphocytes, and NK lymphocytes via flow cytometry, ELISA, ELISPOT, immunoblot, and microarray assays.
  Other Names: Correlatives studies; laboratory biomarker analysis

SUMMARY:
This research trial studies lymphocyte profiles and activation status in patients with graft-versus-host disease. Studying samples of blood in the laboratory from patients with cancer may help doctors identify and learn more about biomarkers related to graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore and assess changes in subsets and activation status of B-, T,-, and natural killer (NK) lymphocytes in peripheral blood following allogeneic stem cell transplant and how they may be associated with clinical events with an ultimate future goal of conducting a larger successor study to identify potential therapeutic targets based on its findings.

SECONDARY OBJECTIVES:

I. To assess the feasibility of obtaining and comparing patients with chronic graft-versus-host disease (cGVHD) with time-matched stem cell transplant (SCT) patients without cGVHD and identify logistical challenges with obtaining and processing samples in each of the subgroups of interest for these analyses.

II. To assess and explore differences in lymphocyte subsets (B-, T-, and NK) between those with vs. without cGVHD.

III. To assess and explore differences in cytokines in patients with cGVHD vs. those without.

IV. To describe lymphocyte subsets and activation and explore how these may be related to specific clinical manifestations of cGVHD.

OUTLINE:

Blood samples are analyzed for activation status of B lymphocytes, T lymphocytes, and NK lymphocytes via flow cytometry, enzyme-linked immunosorbent assay (ELISA), enzyme-linked immunosorbent spot (ELISPOT), immunoblot, and microarray assays.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic SCT groups: Patients who have received stem cell transplantation at The Ohio State University are eligible and who are at or beyond day +75 following allogeneic SCT regardless of previous diagnosis of acute or chronic graft-versus-host disease (GVHD)
* Autologous SCT group: Patients who have received an autologous stem cell transplant at The Ohio State University and who have achieved platelet and neutrophil engraftment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received an autologous stem cell transplant and stem cell transplant at The Ohio State University.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Subsets and activation status of B, T, and NK lymphocytes | Up to 2 months
  Side by side box plots with overlaid plotted points will be used to assess potential differences in continuous markers between groups.

SECONDARY OUTCOMES:
Logistical challenges with obtaining and processing samples in each of the subgroups of interest | Up to 2 months
Differences in lymphocyte subsets (B, T, and NK) between those with vs. without cGVHD | Up to 2 months
Differences in cytokines in patients with cGVHD vs. those without | Up to 2 months
Differences in in lymphocyte activation between those with vs. without cGVHD | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Jaglowski, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu